CLINICAL TRIAL: NCT06397638
Title: Rescue Carotid Stenting in Tandem Occlusions: 4-year Experience From a Comprehensive Stroke Centre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Can Tho Stroke International Services Hospital (Other)
Responsible Party: Principal Investigator, Dr. Cuong Tran Chi, Director - Doctor, Can Tho Stroke International Services Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Rescue carotid stenting
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Acute Stroke; Ischemic Stroke, Acute
Keywords: tandem occlusions; rescue carotid stenting; anterior circulation
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rescue carotid stenting (Experimental): Rescue carotid stenting in tandem occlusions
  Interventions: Procedure: Rescue carotid stenting

INTERVENTIONS:
Procedure: Rescue carotid stenting — Rescue carotid stenting in tandem occlusions

SUMMARY:
The rescue carotid stenting has recently been an additional treatment followed by mechanical thrombectomy in tandem occlusions of the anterior circulation. Nevertheless, there were few data to date that support this beneficial treatment in Asia. The investigators hypothesized that this treatment related to improvement of clinical outcomes after procedure.

DETAILED DESCRIPTION:
The anterior circulation made commonly up 70-80% of all ischemic strokes. The mechanical thrombectomy is the gold treatment standard in acute ischemic stroke due to large vessel occlusion of anterior circulation. Tandem occlusions are one of the acute lesions relating to the high poor clinical outcome rate. Besides, tandem characteristic is a challenge to perform endovascular therapy and save procedural time in the restoration blood flow to the cerebral artery territory infarction. Many studies demonstrated the roles of rescue carotid stenting with either proximal-to-distal or distal-to-proximal approach in the successful recanalization of tandem occlusions. However, few studies analyzed in detail this beneficial treatment in Asia. Therefore, the investigators conducted this study to assess whether rescue carotid stenting in the tandem occlusions to improve clinical outcomes at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Onset to treatment time < 24 hours
* NIHSS > 5
* DWI-ASPECTS ≥ 5

Exclusion Criteria:

* Premorbid mRS > 2
* Loss to follow-up after discharge

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
The good 3-month outcome rate | 3 months
  The good 3-month outcome rate was accessed by modified Rankin Score (mRS ≤ 2).

CONTACTS AND LOCATIONS:
Overall Officials: Cuong C Tran, PhD, Principal Investigator — Can Tho Stroke International Services General Hospital
Locations (1):
- Can Tho SIS Hospital, Can Tho, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allard J, Delvoye F, Pop R, Labreuche J, Maier B, Marnat G, Sibon I, Zhu F, Lapergue B, Consoli A, Spelle L, Denier C, Richard S, Piotin M, Gory B, Mazighi M; ETIS Investigators. 24-Hour Carotid Stent Patency and Outcomes After Endovascular Therapy: A Multicenter Study. Stroke. 2023 Jan;54(1):124-131. doi: 10.1161/STROKEAHA.122.039797. Epub 2022 Dec 21. PMID 36542074
- [Background] Zevallos CB, Farooqui M, Quispe-Orozco D, Mendez-Ruiz A, Dajles A, Garg A, Galecio-Castillo M, Patterson M, Zaidat O, Ortega-Gutierrez S. Acute Carotid Artery Stenting Versus Balloon Angioplasty for Tandem Occlusions: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2022 Jan 18;11(2):e022335. doi: 10.1161/JAHA.121.022335. Epub 2022 Jan 13. PMID 35023353
- [Background] Anadani M, Marnat G, Consoli A, Papanagiotou P, Nogueira RG, Siddiqui A, Ribo M, Spiotta AM, Bourcier R, Kyheng M, Labreuche J, de Havenon A, Sibon I, Dargazanli C, Arquizan C, Cognard C, Olivot JM, Anxionnat R, Audibert G, Mazighi M, Blanc R, Lapergue B, Richard S, Gory B; TITAN and ETIS Registry Investigators. Endovascular Therapy of Anterior Circulation Tandem Occlusions: Pooled Analysis From the TITAN and ETIS Registries. Stroke. 2021 Oct;52(10):3097-3105. doi: 10.1161/STROKEAHA.120.033032. Epub 2021 Aug 10. PMID 34372671